CLINICAL TRIAL: NCT01903174
Title: AeroForm Patient Controlled Tissue Expansion for Breast Reconstruction
Brief Title: Study of AeroForm Tissue Expander for Breast Reconstruction
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AirXpanders, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-0004
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer; Breast Reconstruction
Keywords: Breast Cancer; Breast Reconstruction; Breast Tissue Expansion; Breast Tissue Expander; Two Stage Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AeroForm Tissue Expansion (Experimental): AeroForm Breast Tissue Expander placed after mastectomy
  Interventions: Device: AeroForm Breast Tissue Expander

INTERVENTIONS:
Device: AeroForm Breast Tissue Expander — Breast Tissue Expander using a remote control to fill the expander with Carbon Dioxide
  Other Names: AeroForm; AeroForm Tissue Expander; AirXpander; AirXpander Tissue Expander; AirXpanders Breast Tissue Expander

SUMMARY:
This study is intended to support previous positive results of the AeroForm™ Patient Controlled Tissue Expander System for breast reconstruction

DETAILED DESCRIPTION:
The objective of this study is to provide performance and safety data to support the clinical use of the AeroForm™ Patient Controlled Tissue Expander System for breast reconstruction in a patient population with a broad selection criteria

ELIGIBILITY:
Inclusion Criteria:

1. Subject is female between the ages of 18 - 70.
2. Subject has elected two stage breast reconstruction with tissue expanders.
3. Subject's tissue is amenable to tissue expansion.
4. Subject is able to provide written informed consent.
5. Subject is able and willing to comply with all of the study requirements.
6. Subject has the physical, perceptual and cognitive capacity to understand and manage the at home dosing regimen.

Exclusion Criteria:

1. Subject has residual gross malignancy following mastectomy.
2. Subject has a current infection at the intended expansion site.
3. Subject has clinically significant radiation fibrosis at the expansion site.
4. Subject has planned radiation at the intended expansion site during the time the expander is implanted.
5. Subject has any co-morbid condition determined by the Investigator to place the subject at an increased risk of complications (e.g., severe collagen vascular disease, poorly managed diabetes).
6. Subject is currently participating in a concurrent investigational drug or device study.
7. Subject is a current tobacco smoker.
8. Subject is overweight with a BMI > 33.
9. Subject has currently implanted electronic device such as a pacemaker, defibrillator, neurostimulator device, or drug infusion device.
10. Subject is pregnant or planning to become pregnant during the study period.
11. Subject has a history of psychological condition, drug or alcohol misuse which may interfere with their ability to use the device safely.

    -

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Successful Tissue Expansion and Exchange to Permanent Breast Implant unless Precluded by a Non-Device Related Event | 6 months

SECONDARY OUTCOMES:
Adverse Events related to the Breast Reconstruction Procedure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tony Connell, F.R.A.C.S., Principal Investigator — Mount Hospital
Locations (1):
- Mount Hospital, Subiaco, Western Australia, Australia